CLINICAL TRIAL: NCT02785471
Title: Assessing Online Interventions for Men's' Mental Health and Wellbeing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: University of Utah (Other)
Responsible Party: Principal Investigator, Jodi Jacobson Frey, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HP-00066262
Record Dates: First submitted 2016-04-06; First posted 2016-05-27 (Estimated); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Mental Health Wellness 1
Keywords: Suicide prevention; men's mental health; depression; suicide ideation and behaviors
MeSH Terms: conditions — Suicide Prevention; Depression; Behavior | interventions — Mass Screening; Mental Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Screening for Mental Health only (Active Comparator): Participants in the Screening for Mental Health only (control) group will complete the online depression and suicide screening and receive immediate feedback and referrals.
  Interventions: Behavioral: Screening for Mental Health only
- Screening for Mental Health & Man Therapy (Experimental): Participants assigned to Screening for Mental Health & Man Therapy (intervention) group will be offered the Man Therapy program in conjunction with Screening for Mental Health.
  Interventions: Behavioral: Screening for Mental Health & Man Therapy

INTERVENTIONS:
Behavioral: Screening for Mental Health only — Participants in the Screening for Mental Health (SMH)-only group will complete the online depression and suicide screening and receive immediate feedback and referrals.
  Arms: Screening for Mental Health only
Behavioral: Screening for Mental Health & Man Therapy — Participants assigned to Screening for Mental Health, plus Man Therapy (SMH+MT) group will be offered the Man Therapy program in conjunction with Screening for Mental Health. MT provides online early intervention services designed specifically for men who are at risk for suicide and are less likely to engage in help-seeking behavior. MT takes an innovative and humorous approach to mental health education and help seeking through a fictional "therapist" named Dr. Rich Mahogany, who is a no-nonsense "man's man" who informs men about the importance of honest talk about life's challenges in addressing their problems. The web portal allows review "manly mental health information, facts and tips," explore "man therapies," and view videos of men with lived experience.
  Arms: Screening for Mental Health & Man Therapy

SUMMARY:
The purpose of this study is to test a comprehensive, male-oriented, online screening and referral (Screening for Mental Health; SMH) and male-oriented online information and referral intervention program (Man Therapy; MT) to improve mental health and wellbeing with a focus on prevention of suicide and help-seeking behaviors among middle-aged men. The online programs will be offered together to maximize the effect on reducing suicide behavior and increasing mental health help-seeking behaviors for men. If successful in decreasing suicide behavior and ideation and increasing suicide help-seeking behavior, this intervention could be scaled up to contribute to a reduction in suicide behaviors and deaths across the country.

ELIGIBILITY:
Inclusion Criteria:

1. men living in Michigan;
2. 25-64 years of age at time of enrollment;
3. scoring in the moderate- to high-risk range (or answering positively on Question 9) on the Harvard Department of Psychiatry/NDSD Scale (HANDS), scoring in the moderate- to high-risk range for anger on the DSM-5 Level 1 Cross-Cutting Symptom Measure, or identifying any risk for suicide ideation or behavior on the Columbia-Suicide Severity Rating Sale (C-SSRS); and
4. fluent in reading English

Exclusion Criteria:

1. females
2. scoring in the low risk range on the Harvard Department of Psychiatry/NDSD Scale (HANDS), scoring in the low risk range for anger on the DSM-5 Level 1 Cross-Cutting Symptom Measure, or not identifying any risk for suicide ideation or behavior on the Columbia-Suicide Severity Rating Sale (C-SSRS); and
3. not fluent in reading English

Ages: 25 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 554 (Actual)
Dates: Start 2016-09; Primary Completion 2019-05-30 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change in depression symptoms as measured by The HANDS: Harvard Department of Psychiatry National Depression Screening Day Scale | Baseline; 2 weeks post randomization; 12 weeks post randomization
Change in suicide risk as measured by the Columbia-Suicide Severity Rating Scale-Screen Version | Baseline; 2 weeks post randomization; 12 weeks post randomization

SECONDARY OUTCOMES:
change in attitudes toward help-seeking behavior as measured by the Attitudes Toward Seeking Professional Help short-form | 2 weeks post randomization; 12 weeks post randomization
change in alcohol use/abuse as measured by the Alcohol Use Disorders Identification Test | 2 weeks post randomization; 12 weeks post randomization
change in relationship conflicts as measured by the Psychological Aggression Scale | 2 weeks post randomization; 12 weeks post randomization
change in financial situation as measured by two items (J1 and J4) of the 2009 National Financial Capability Study, Financial Industry Regulatory Authority | 2 weeks post randomization; 12 weeks post randomization
change in social support as measured by the Perceived Social Support and/or Conflict scale | 2 weeks post randomization; 12 weeks post randomization
change in interpersonal needs as measured by the Interpersonal Needs Questionnaire | 2 weeks post randomization; 12 weeks post randomization
change in drug use/abuse as measured by the National Institute of Drug Abuse Quick Screen | 2 weeks post randomization; 12 weeks post randomization
change in physical aggression as measured by the Physical Aggression Index scale | 2 weeks post randomization; 12 weeks post randomization
change in help seeking behavior as measured by the Perceived Stigma and Barriers to Care for Psychological Problems scale | 2 weeks post randomization; 12 weeks post randomization
change in help seeking behavior as measured by the General Help Seeking Questionnaire | 2 weeks post randomization; 12 weeks post randomization
change in physical and mental health as measured by the Healthy Days Measures | 2 weeks post randomization; 12 weeks post randomization
change in anger as measures by the DSM-5 Self Rated Level 1 Cross-Cutting Symptom Measure | Baseline; 2 weeks post randomization; 12 weeks post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Jodi Jacobson Frey, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gilgoff JN, Wagner F, Frey JJ, Osteen PJ. Help-seeking and Man Therapy: The impact of an online suicide intervention. Suicide Life Threat Behav. 2023 Feb;53(1):154-162. doi: 10.1111/sltb.12929. Epub 2022 Nov 22. PMID 36412229
- [Derived] Frey JJ, Osteen PJ, Sharpe TL, Mosby AO, Joiner T, Ahmedani B, Iwamoto D, Nam B, Spencer-Thomas S, Ko J, Ware OD, Imboden R, Cornette MM, Gilgoff J. Effectiveness of man therapy to reduce suicidal ideation and depression among working-age men: A randomized controlled trial. Suicide Life Threat Behav. 2023 Feb;53(1):137-153. doi: 10.1111/sltb.12932. Epub 2022 Nov 14. PMID 36373571